CLINICAL TRIAL: NCT04288011
Title: Validation of the BeCare Multiple Sclerosis Assessment App
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BeCare Link LLC (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000023992
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
Keywords: MS; mobile app; machine learning; EDSS; BeCare
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical EDSS: The Kurtzke EDSS, is a clinical rating scale for multiple sclerosis having scores between 0 to 10 that are assigned by a trained clinician. Smaller impairments are assessed at lower scores and disability is assessed at higher scores. It is important to note, however, that despite being denoted on an ordinal scale, each level on the scale is not indicative of an equal change in disability.
- MLA EDSS: The Kurtzke EDSS, is a clinical rating scale or multiple sclerosis having scores between 0 to 10 that are assigned by a technique based upon several different Machine Learning Algorithms that are combined to produce a single score

SUMMARY:
This study involves data collection from use of the BeCare Link LLC mobile device app by subjects with Multiple Sclerosis.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study over a period of 12 months beginning at the time of IRB approval or until a complete data set is collected on 50 subjects. This will be a longitudinal study following individual patients for six months and data collection for all patients will continue for a total of 18 months. Patients will be enrolled during their first visit. Additionally, at the first visit for each patient, an EDSS score will be measured, app training performed, and the first app-obtained measurements entered. The patients will be contacted by the research assistant to complete the app tasks on a weekly basis. Clinical EDSS scores will be measured in the clinic at 3 month and 6 month follow-up appointments Research personnel at the Clinical Site will screen for eligible subjects and obtain informed consent. The data collected from the application will continue to be sent to the sponsor.

The purpose of the BeCare App is to replicate the clinically-derived EDSS score. Because the app can be used independently by the patients at more frequent intervals, use of the app may lead to earlier detection of a decline in function than would be possible by clinic evaluations; the app would measure function utilizing data that closely parallels the clinically obtained EDSS score. In the clinic it may take up to two years before someone is noted to have progressive features. The implication of using the BeCare MS App is earlier intervention with switching to more effective Disease Modifying Treatment. Further, as the BeCare App has a cognitive assessment component not routinely performed during follow-up clinical visits, the need for earlier intervention may result in more effective therapy and, therefore, slowed disease progression.

The EDSS is scored by first assessing Human Functional systems (FS) scores. These systems include Sensory, Bowel& Bladder, Cerebral, Ambulation and Visual. Function System Scores correspond to the amount of observed disability in that system. Low scores 0 represent no disability in that system, to a maximum score representing high disability.

Clinicians then assess EDSS scores from these Functional System scores (FS) according to their experience with patients. The EDSS is scored according to the following:

0 Normal neurological exam, no disability in any FS 1.0 No disability, minimal signs in one FS 1.5 No disability, minimal signs in more than one FS 2.0 Minimal disability in one FS 2.5 Mild disability in one FS or minimal disability in two FS 3.0 Moderate disability in one FS, or mild disability in three or four FS. No impairment to walking 3.5 Moderate disability in one FS and more than minimal disability in several others. No impairment to walking 4.0 Significant disability but self-sufficient and up and about some 12 hours a day. Able to walk without aid or rest for 500m 4.5 Significant disability but up and about much of the day, able to work a full day, may otherwise have some limitation of full activity or require minimal assistance. Able to walk without aid or rest for 300m 5.0 Disability severe enough to impair full daily activities and ability to work a full day without special provisions. Able to walk without aid or rest for 200m 5.5 Disability severe enough to preclude full daily activities. Able to walk without aid or rest for 100m 6.0 Requires a walking aid - cane, crutch, etc. - to walk about 100m with or without resting 6.5 Requires two walking aids - pair of canes, crutches, etc. - to walk about 20m without resting 7.0 Unable to walk beyond approximately 5m even with aid. Essentially restricted to wheelchair; though wheels self in standard wheelchair and transfers alone. Up and about in wheelchair some 12 hours a day 7.5 Unable to take more than a few steps. Restricted to wheelchair and may need aid in transferring. Can wheel self but cannot carry on in standard wheelchair for a full day and may require a motorised wheelchair 8.0 Essentially restricted to bed or chair or pushed in wheelchair. May be out of bed itself much of the day. Retains many self-care functions. Generally has effective use of arms 8.5 Essentially restricted to bed much of day. Has some effective use of arms retains some self-care functions 9.0 Confined to bed. Can still communicate and eat 9.5 Confined to bed and totally dependent. Unable to communicate effectively or eat/swallow 10.0 Death due to MS

ELIGIBILITY:
Inclusion Criteria:

1. A history of Multiple Sclerosis, which will be verified through medical records and will be classified as clinically definite based on revised McDonald criteria
2. Between the ages 18-75
3. Mild to moderate disability in one or more of the modalities assessed by the BeCare App.
4. Ability to provide Informed Consent.

Exclusion Criteria:

1. Subjects at risk of falling
2. Subjects with poor vision that cannot read the screen of a mobile phone

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate Multiple Sclerosis that can use a mobile app and are ambulatory.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Clinical EDSS score vs MLA EDSS score comparison | day 1 (initial visit)
  To assess the efficacy of using a mobile application to perform routine assessments of neurological and physical functioning in subjects with MS by comparing clinically assigned EDSS scores with EDSS scores assigned by a single or multiple artificial intelligence techniques at various timed intervals
Clinical EDSS score vs MLA EDSS score comparison | 90 days after day 1
  To assess the efficacy of using a mobile application to perform routine assessments of neurological and physical functioning in subjects with MS by comparing clinically assigned EDSS scores with EDSS scores assigned by a single or multiple artificial intelligence techniques at various timed intervals
Clinical EDSS score vs MLA EDSS score comparison | 180 days after day 1
  To assess the efficacy of using a mobile application to perform routine assessments of neurological and physical functioning in subjects with MS by comparing clinically assigned EDSS scores with EDSS scores assigned by a single or multiple artificial intelligence techniques at various timed intervals

SECONDARY OUTCOMES:
Disease Progression Measured by Change in EDSS score | weekly for 26 weeks
  To improve the understanding of disease progression over a shorter time interval captured by weekly BeCare application's monitoring.
Development of a novel application to measure change in MS | 18 months
  To assist in the development of a novel application that is easy to use and is capable of evaluating MS patients' neurological and physical functioning outside the clinical setting, that allows both patients and clinicians to view their disease progression over time. The data this application will collect could prove to be a valuable source of information and may improve how well MS symptoms and functioning can be evaluated by healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Stoll, DO,MS, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] Berrigan LI, Fisk JD, Walker LA, Wojtowicz M, Rees LM, Freedman MS, Marrie RA. Reliability of regression-based normative data for the oral symbol digit modalities test: an evaluation of demographic influences, construct validity, and impairment classification rates in multiple sclerosis samples. Clin Neuropsychol. 2014;28(2):281-99. doi: 10.1080/13854046.2013.871337. Epub 2014 Jan 20. PMID 24438521